CLINICAL TRIAL: NCT01026428
Title: A Randomised, Double-blind, Placebo-controlled, Two-period, Two-sequence-crossover Interaction Study to Assess the Effect of Safinamide on Levodopa Pharmacokinetics in Subjects With Parkinson's Disease
Brief Title: A Study to Assess the Effect of Safinamide on Levodopa Pharmacokinetics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 28780
Record Dates: First submitted 2009-12-01; First posted 2009-12-04 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-01

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: safinamide; levodopa; drug -drug interaction; pharmacokinetics; Patients diagnosed with idiopathic Parkinson's disease, levodopa-responsive, treated with a stable dose of levodopa/carbidopa
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safinamide + Levodopa (Experimental)
  Interventions: Drug: Safinamide + Levodopa
- Placebo + Levodopa (Placebo Comparator)
  Interventions: Other: Placebo + Levodopa

INTERVENTIONS:
Drug: Safinamide + Levodopa — Treatment A: 100mg safinamide once daily administration for 6 days + immediate release levodopa formulation (100 mg levodopa + 25 mg carbidopa = Nacom®).
  Arms: Safinamide + Levodopa
Other: Placebo + Levodopa — Treatment B: Placebo matching 100mg safinamide once daily administration for 6 days + immediate release levodopa formulation (100 mg levodopa + 25 mg carbidopa = Nacom®).
  Arms: Placebo + Levodopa

SUMMARY:
The objective of this study is to investigate the effect of safinamide on levodopa blood levels, both after single and multiple dosing of safinamide . A further objective of the study is to assess the safety and tolerability of safinamide when given together with levodopa in the applied regimen.

For that purpose, all study participants will undergo intensive blood sampling for investigation of levodopa levels and various tolerability examinations, such as the measurement of vital signs (blood pressure, pulse, body temperature), recording of ECGs and questioning to find out how the study participants are feeling. Furthermore, blood samples will be drawn and urine tests will be performed repeatedly for safety purpose during the course of the study.

The results of this clinical trial may be used for the drug registration of safinamide in the future.

DETAILED DESCRIPTION:
Treatments are given in a crossover design.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: male or female
2. Age: 30 years
3. Body Mass Index (BMI): 18 - 32 kg/m2
4. Diagnosed with idiopathic Parkinson's disease, with Hoehn and Yahr (H&Y) of I-III
5. Levodopa-responsive patients treated with a stable dose of levodopa/carbidopa
6. Electrocardiogram recording (12 leads) normal or with abnormalities which are not hazardous to the patient according to the opinion of the investigator.
7. Negative beta-HCG test and not lactating (females). Women who are of childbearing potential must be using acceptable methods of contraception and should be informed of the potential risks associated with becoming pregnant while enrolled within a clinical research study. Accepted forms of contraception are: i.e. intrauterine device and a barrier method, combined oral contraceptives and a barrier method, or double-barrier method throughout the study. Female volunteers who are post -menopausal or surgically sterile may be enrolled
8. Ability to maintain an accurate and complete dosing diary, with the help of a caregiver, recording doses of levodopa and study medication taken at home All parameters will be determined within three weeks prior to first dosing. Subjects must have given written informed consent before any study-related activities are carried out

Exclusion Criteria:

To be eligible for inclusion in this study the subjects must not meet any of the following criteria:

1. Co-administration of other drugs causing dopamine release (e.g. reserpine) or affecting levodopa metabolism (e.g COMT inhibitors except AADC inhibitors) or any other medication clinically contraindicated with MAO B inhibitors or with levodopa/carbidopa Note: Use of Selective serotonin reuptake inhibitors [SSRI] and selective noradrenalin reuptake inhibitors [SNRI] will be permitted, provided the dose is kept as low as possible and remains stable throughout the trial.
2. Co-administration of other MAO inhibitors (e.g. selegiline, rasagiline)
3. The patient is in a late stage of Parkinson's disease, and is experiencing severe, disabling peak-dose or biphasic dyskinesia and/or unpredictable or widely swinging fluctuations in their symptoms
4. Any indication of forms of Parkinsonism, other than idiopathic Parkinson's disease.
5. Treatment with any agent known to inhibit or induce drug-metabolizing enzymes (e.g., barbiturates, St John's Wort etc.) within 4 weeks prior study treatment
6. Concomitant oral iron treatment
7. History of hypersensitivity or contraindications to MAO-B inhibitors or levodopa
8. Clinically relevant allergies (especially hypersensitivity toward any medicinal drugs)
9. Significant hepatic impairment
10. Significant renal impairment
11. Diseases or surgeries of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility
12. Diagnosis of Human Immunodeficiency Virus (HIV), or acute Hepatitis B or C
13. Clinically relevant disease which in the investigator's opinion would exclude the subject from the study, such as significant cardiovascular and lung diseases, narrow-angle glaucoma or endocrinological diseases such as hyperthyroidism or pheochromocytoma
14. A neoplastic disorder, which is either currently active or has been in remission for less than one year.
15. Active psychiatric disease (e.g, schizophrenia, psychotic depression)
16. History of melanoma or current cancer disease and undiagnosed, but melanoma suspicious skin lesion
17. Signs for dementia which could interfere with the compliance to the study as judged by the investigator
18. Ophthalmologic history including any of the following conditions: albino subjects, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity (i.e., 20/70), retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation (uveitis), or diabetic retinopathy.
19. Consumption of important quantities of coffee or tea corresponding to more than 600 mg caffeine/day, or tobacco smoking (more than 10 cigarettes per day)
20. Diet considerably deviating from normal nutritional patterns (e.g. vegan; diets with very high protein content [Atkins])
21. Participation in another clinical study within 30 days prior to the planned first drug administration
22. Alcohol and drug abuse (during the past three years)
23. Transfusion of blood or plasma derivatives within 3 month prior to the planned first drug administration
24. Blood donation within 90 days before the start of the clinical study
25. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
AUC and Cmax of Levodopa | Main pharmacocinetics measurements will be taken at Day 1 and 6 of each period.

SECONDARY OUTCOMES:
tmax, CL, t1/2 of Levodopa | Main pharmacocinetics measurements will be taken at Day 1 and 6 of each period.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Krösser, PhD, Study Director — Merck KGaA, Darmstadt, Germany
Locations (2):
- Italy (2):
  - Research Site, Casino
  - Research Site, Roma